

## CLINICAL TRIAL PROTOCOL

# Investigational Product: UBITh® CGRP Immunotherapy (UB-313)

A Phase 1 Randomized, Double-Blind, Placebo-Controlled, First-in-Human Study to Evaluate the Safety, Tolerability, and Immunogenicity of UBITh® CGRP Immunotherapy (UB-313) in Healthy Participants

EudraCT: 2022-000798-19

Protocol Number: Final Version 3.0
UB-313-101 Date: 13 APRIL 2023

This document contains confidential information and is the property of Vaxxinity Ltd. (Vaxxinity, further referred to as the Sponsor). The receiver(s) of this document understand(s) and agree(s) that this document is not to be disclosed to any unauthorized third party without prior written agreement issued by the Sponsor. The need to disclose certain information contained in this document for the purpose of obtaining informed consent from potential participants or their legally acceptable representative(s) will be considered as exceptions.



# **SYNOPSIS**

| Protocol Number | UB-313-101 |
|---|---|
| Title of Study | A Phase 1 Randomized, Double-Blind, PlaceboControlled, First-in-Human Study to Evaluate the Safety, Tolerability, and Immunogenicity of UBITh® CGRP Immunotherapy (UB-313) in Healthy Adults |
| Study Site | This study will be conducted at one study center (Center for Clinical Pharmacology) in Leuven, Belgium |
| <b>Development Phase</b> | Phase 1, First-in-human |
| Study Objectives | <ul> <li>Primary Objectives:</li> <li>To evaluate the safety and tolerability of UB-313, when administered at selected dose regimens given intramuscularly (IM) to healthy adults.</li> <li>To evaluate the anti-calcitonin gene-related peptide (anti-CGRP) specific antibody responses to selected UB-313 dose regimens in healthy adults.</li> </ul> |
| | Secondary Objective: To evaluate the effects of selected UB-313 dose regimens on capsaicin-induced dermal blood flow (DBF) as a surrogate marker of target engagement. |
| | <ul> <li>Exploratory Objectives:</li> <li>To evaluate the effects of selected UB-313 dose regimens on CGRP concentrations in serum.</li> <li>To characterize antibodies generated by UB-313.</li> <li>To examine cytokine release induced by UB-313.</li> </ul> |
| Endpoints | Primary Endpoints Safety will be assessed by adverse events (AEs), adverse events of special interest (AESIs), medically attended adverse events (MAAEs), local (injection site) and systemic (generalized) reactions (i.e., reactogenicity), clinical laboratory assessments (e.g., chemistry, hematology, urinalysis), vital signs, neurological and physical examinations, and electrocardiograms (ECGs) through the end of study. Immunogenicity will be measured by serum anti-CGRP antibody titers and analyzed from baseline to Week 16 and through the end of study (Week 44). |
| | Secondary Outcome Measure/Endpoints |
| | Pharmacodynamics (PD) of the immune response will be measured by the inhibition of capsaicin-induced increase in DBF and analyzed from baseline to Week 16 and either until return to baseline <i>or</i> until Week 44, whichever comes first. |
| | Exploratory Outcome Measures/Endpoints |
| | <ul> <li>Exploratory outcome measures may include but are not limited to the following:</li> <li>CGRP concentrations in serum through the end of study.</li> <li>Antibody titers against components of UB-313 (i.e., CpG1 and UBITh1) through the end of study.</li> <li>Isotype-specific anti-CGRP antibody titers through the end of study.</li> <li>Cytokine release from peripheral blood mononuclear cells stimulated with a component of UB-313 (T-cell ELISpot) through Week 16.</li> </ul> |



#### Methodology

This single center, double-blind, placebo-controlled, multidose regimen, first-in-human (FIH) study of UB-313, an anti-CGRP peptide -based immunotherapeutic candidate, is designed to assess the safety, tolerability, and immunogenicity of 4 selected UB-313 dose regimens in healthy adults.

#### **Screening Period**

All participants will undergo Laser Speckle Contrast Imaging (LSCI) assessments at Screening to ensure a capsaicin response of at least 100% increase in DBF.

Following Screening, all eligible participants (approximately 40) will be randomized to receive 3 IM injections of UB-313 or placebo in a staggered manner by cohort as described below.

#### **Investigational Product Dosage and Schedule:**

| Cohort | Number of Participants | Dose Regimen (0.5mL) | | |
|---|---|---|---|---|
| | | Week 1 | Week 4 | Week 12 |
| 1 | 8 | 100 μg | 100 μg | 100 μg |
| (N=10) | 2 | Placebo | Placebo | Placebo |
| 2 | 8 | 300 μg | 100 μg | 100 μg |
| (N=10) | 2 | Placebo | Placebo | Placebo |
| 3 | 8 | 300 μg | 300 μg | 300 μg |
| (N=10) | 2 | Placebo | Placebo | Placebo |
| 4 | 8 | 600 μg | 100 μg | 100 μg |
| (N=10) | 2 | Placebo | Placebo | Placebo |

### **Double-Blind Period**

Eligible healthy participants will be enrolled into 1 of the 4 cohorts, as previously described. For safety purposes, dosing of all cohorts will be staggered. Sentinel dosing will be performed in Cohorts 1 (first dose of 100  $\mu g$ ), 2 (first dose of 300  $\mu g$ ), and 4 (first dose of 600  $\mu g$ ). The remaining participants in a cohort may be enrolled following a safety review conducted at least 24-hours after sentinel dosing; however, no more than 4 participants will be dosed within a 24-hour period.

Once all escalation safety evaluable participants within each of the dose levels (100  $\mu g$  for Cohort 1, and 300  $\mu g$  in Cohorts 2 and 3) have been observed for 1 week following their first dose of study Investigational Medicinal Product (IMP), all available safety data will be reviewed by the Safety Review Committee (SRC) before progressing to the next higher dose cohort (100  $\mu g$  to 300  $\mu g$  to 600  $\mu g$ ).



| | Cohort 3 may begin dosing at least 24 hours after all participants in Cohort 2 have received their first dose, and available (blinded) safety and tolerability data have been reviewed by the SRC. Based on the available data, a decision will be made to begin dosing of Cohort 3. Participants will be provided with a diary. Starting the day of IMP administration, they will fill in the diary daily for 7 days, recording their |
|---|---|
| | temperature, and any solicited local and systemic symptoms of reactogenicity. |
| | Capsaicin Challenge |
| | A capsaicin-induced increase in DBF model will be used to assess the PDs of the UB-313-mediated immune response. Personnel who will perform these assessments will not be involved in UB-313 safety and tolerability evaluation due to the potential of unblinding. The capsaicin challenge will be conducted at Screening, Baseline before the first dose, and every 4 weeks up to Week 20 and subsequently every 8 weeks until the end of study at Week 44. After Week 16, LSCI assessment may no longer be required once the average capsaicin induced DBF increase within that cohort has returned to baseline (i.e., DBF response ±2 SD before administration of IMP within a cohort). |
| Total Expected Number of Participants | Approximately 40 eligible healthy male and female participants (10 per cohort) will be enrolled to receive UB-313 or placebo. |
| Main Inclusion Criteria | <ul> <li>Full details of inclusion criteria are listed in the protocol. The main inclusion criteria include:</li> <li>Is a male or female aged 18 to 55 years old, inclusive, at time of informed consent.</li> <li>Has a body mass index between 18 and 30 kg/m², inclusive at Screening, and with a minimum weight of 50 kg.</li> <li>Male participants and their partners of childbearing potential must commit to the use of highly effective contraceptives for the study duration and for at least 12 weeks after the last dose. Men must refrain from donating sperm during this same period.</li> <li>Female participants must be of nonchildbearing potential, or, for women of childbearing potential, must be willing to practice highly effective contraception throughout the duration of the study and for at least 24 weeks following the last dose.</li> </ul> |
| Main Exclusion Criteria | Full details of exclusion criteria are listed in the protocol. The main exclusion criteria include: • Has a history of clinically significant medical or psychiatric conditions, |
| | which in the opinion of the Investigator may compromise the participant's safety or the scientific value of the study, posing an unacceptable risk to the participant or interfere with the participant's ability to comply with study procedures or abide by study restrictions. |
| | Presents any concern by the Investigator regarding safe participation in the study or for any other reason (including contraindication to MRI) that the Investigator considers the participant inappropriate for participation in the study. Has a recent history (within the past year of Screening) of migraine. |
| | Has a recent history (within the past year of Screening) of migraine headache. |
| | Has unsuitable skin characteristics for the dermal capsaicin challenge as determined by the Investigator. |



| | Has not demonstrated at least a 100% increase in DBF following capsaicin challenge as part of Screening procedures and measured through LSCI. |
|---|---|
| Investigational Medicinal<br>Product | UB-313 drug product is a synthetic CGRP peptide-based immunotherapy formulated in CpG1 and Adju-Phos <sup>®</sup> . It is provided in single dose vial (peptide: 100 μg, 300 μg, or 600 μg; dosage volume: 0.5 mL). |
| | <b>Placebo</b> is 0.9% sodium chloride (normal saline), preservative free for injection. |
| | IMP will be either UB-313 or placebo and can also be referred to as study drug. |
| Participation Duration | The total study participation will last up to 48 weeks, including: Screening period: up to 4 weeks Double-blind period: 44 weeks |
| Statistical Considerations | As this is an FIH study, the sample size is based on the exploratory nature of the design. No statistical power to be considered to determine the sample size. Primary time-points for immunogenicity and PD are two-fold: a) First phase at the end of Week 16 for evaluating maximal immuno-responses elicited by the 4 dosage regimens (i.e., cohorts) of UB-313 b) Second phase of response maintenance period after Week 16 until the end of study (Week 44), in which effects of the 4 dosage regimens of UB-313 on the duration of responses will be evaluated. When any cohort completes Week 16, first phase analyses can be conducted based on cleaned cohort data up to Week 16. To maintain blinding for the remainder of the study, the first phase analyses will be conducted and reviewed only by a designated and independent team before the end of study final database lock. The purpose of the early analyses of first phase data prior to the completion of the study is to have an early read out of the first part of the primary immunogenicity and PD results to refine the development plan. Design of the second phase of the study will not be changed based on results from the first phase data. |



# **Table 1:** Study Schedule of Assessments

The Investigator may perform visits outside of the scheduled study visits (unscheduled visits) listed in the Schedule of Assessments table to conduct evaluations or assessments required to protect the well-being of the participant.

| Visit Number <sup>1</sup> | Screen <sup>2</sup> | V1 | [2,5 | V1a <sup>5</sup> | V1b <sup>5</sup> | V2 | V | 735 | V3a <sup>5</sup> | V3b <sup>5</sup> | V4 | V5 | V6 <sup>5</sup> | | V6a <sup>5</sup> | V6b <sup>5</sup> | V7 | V8 | V9,<br>V10,<br>V11 | V12/ET |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | Up to 4<br>wks | | W | | | W1 | W4 | | | W5 | W8 | | W12 | | | W13 | W16 | W20,<br>W28,<br>W36 | W44 | |
| Day (Visit<br>Window) | -28 to -<br>1 | D1<br>(-3D) | D1<br> | D2 | D3 | D8<br>(±3D) | D29<br>(-3D) | D29<br>(±3D) | D30 | D31 | D36<br>(±3D) | D57<br>(±5D) | D85<br>(-3D) | D85<br>(±3D) | D86 | D87 | D92<br>(±3D) | D113<br>(±7D) | D141,<br>D197,<br>D253<br>(±14D) | D309<br>(±14D) |
| Visit Type | SRN | Pre<br>IMP | IMP | CRU | TC | CRU | Pre<br>IMP | IMP | CRU | TC | CRU | CRU | Pre<br>IMP | IMP | CRU | TC | CRU | EoT<br>CRU | CRU | EoS/ET<br>CRU |
| General Assessm | ents and Pi | rocedure | S | | | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | | | | |
| Demographic | X | | | | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | | | | |
| Eligibility assessment | X | X | | | | | | | | | | | | | | | | | | |
| Medication review | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| AE/SAE<br>review <sup>3</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Investigational M | ledicinal P | roduct A | dministr | ation an | d Assess | ments | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | | | |
| IMP Injection <sup>18</sup> | | | X | | | | | X | | | | | | X | | | | | | |
| Solicited local<br>and systemic<br>reactions<br>assessment | | | X | | | | | X | | | | | | X | | | | | | |
| Extended unit<br>stay <sup>5</sup> | | | $X^5$ | | | | | X | | | | | | X | | | | | | |
| Diary review <sup>10</sup> | | | X | X | | X | | X | X | | X | | | X | X | | X | | | |
| General Safety A | ssessments | 1 | | | | | • | • | • | | | • | | • | | | • | | | |
| Vital signs (pre-<br>and post-IMP) <sup>6,7</sup> | X | | X | X | | X | | X | X | | X | X | | X | X | | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | | | | |

CONFIDENTIAL Page 6 of 9



| Visit Number <sup>1</sup> | Screen <sup>2</sup> | V1 | V1 <sup>2,5</sup> | | V1b <sup>5</sup> | V2 | \ | 735 | V3a <sup>5</sup> | V3b <sup>5</sup> | | V5 | Vo | 65 | V6a <sup>5</sup> | V6b <sup>5</sup> | V7 | V8 | V9,<br>V10,<br>V11 | V12/ET |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | Up to 4<br>wks | | W | 70 | | W1 | W4 | | | | W5 | W8 | | | | | W16 | W20,<br>W28,<br>W36 | W44 | |
| Day (Visit<br>Window) | -28 to -<br>1 | D1<br>(-3D) | D1<br> | D2 | D3 | D8<br>(±3D) | D29<br>(-3D) | D29<br>(±3D) | D30 | D31 | D36<br>(±3D) | D57<br>(±5D) | D85<br>(-3D) | D85<br>(±3D) | D86 | D87 | D92<br>(±3D) | D113<br>(±7D) | D141,<br>D197,<br>D253<br>(±14D) | D309<br>(±14D) |
| Visit Type | SRN | Pre<br>IMP | IMP | CRU | TC | CRU | Pre<br>IMP | IMP | CRU | TC | CRU | CRU | Pre<br>IMP | IMP | CRU | TC | CRU | EoT<br>CRU | CRU | EoS/ET<br>CRU |
| Weight | X | | X | | | | | X | | | | | | X | | | | X | X | X |
| Physical exam <sup>4,8</sup> | X | | X | | | | | X | | | | | | X | | | | X | | X |
| Neurological<br>exam <sup>4,8</sup> | X | | X | | | | | X | | | | | | X | | | | X | | X |
| Triplicate<br>ECGs <sup>4</sup> | X | | X | | | X | | X | | | X | | | X | | | X | X | X | X |
| MRI <sup>17</sup> | X | | | | | | | | | | | | | | | | | | | |
| Laboratory Asses | ssments4,9 | • | | • | | • | | • | | | • | | • | | • | • | • | • | • | |
| HIV, HCV,<br>HBV | X | | | | | | | | | | | | | | | | | | | |
| Coagulation | X | | | | | | | | | | | | | | | | | | | |
| Clinical<br>chemistry <sup>4</sup> | X | X | | | | X | X | | | | X | X | X | | | | X | X | | X |
| Hematology <sup>4</sup> | X | X | | | | X | X | | | | X | X | X | | | | X | X | | X |
| Urinalysis <sup>4</sup> | X | X | | | | | X | | | | | | X | | | | | X | | X |
| Urine drug<br>screen <sup>4</sup> | X | X | | | | | X | | | | | | X | | | | | | | |
| Pre-IMP<br>alcohol breath<br>test <sup>4</sup> | X | | X | | | | | X | | | | | | X | | | | | | |
| Pre-IMP<br>pregnancy<br>test <sup>4,11</sup> | X | | X | | | | | X | | | | | | X | | | | | | |
| FSH <sup>11</sup> | X | | | | | | | | | | | | | | | | | | | |
| Inflammatory<br>markers <sup>4,12</sup> | X | X | | | | | X | | | | | | X | | | | | X | | X |
| Cytokine panel<br>(pre- and post-<br>IMP) <sup>13</sup> | | X | X | | | | X | X | | | | | X | X | | | | | | |
| Pharmacodynam | ic Assessm | ents <sup>4</sup> | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • |
| Serum<br>antibodies <sup>4,14</sup> | | X | | | | X | X | | | | X | X | X | | | | X | X | X | X |
| Serum CGRP <sup>4</sup> | | X | | | | X | X | | | | X | X | X | | | | X | X | X | X |

CONFIDENTIAL Page 7 of 9



| Visit Number <sup>1</sup> | Screen <sup>2</sup> | V1 | [2,5 | V1a <sup>5</sup> | V1b <sup>5</sup> | V2 | \ | / <b>3</b> <sup>5</sup> | V3a <sup>5</sup> | V3b <sup>5</sup> | V4 | V5 | V6 <sup>5</sup> V6a <sup>5</sup> V6b <sup>5</sup> | | V7 | V8 | V9,<br>V10,<br>V11 | V12/ET | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | Up to 4<br>wks | | V | VO | | W1 | | W | 4 | | W5 | W8 | | W12 | | | W13 | W16 | W20,<br>W28,<br>W36 | W44 |
| Day (Visit<br>Window) | -28 to -<br>1 | D1<br>(-3D) | D1<br> | D2 | D3 | D8<br>(±3D) | D29<br>(-3D) | D29<br>(±3D) | D30 | D31 | D36<br>(±3D) | D57<br>(±5D) | D85<br>(-3D) | D85<br>(±3D) | D86 | D87 | D92<br>(±3D) | D113<br>(±7D) | D141,<br>D197,<br>D253<br>(±14D) | D309<br>(±14D) |
| Visit Type | SRN | Pre<br>IMP | IMP | CRU | TC | CRU | Pre<br>IMP | IMP | CRU | TC | CRU | CRU | Pre<br>IMP | IMP | CRU | TC | CRU | EoT<br>CRU | CRU | EoS/ET<br>CRU |
| PBMC for<br>ELISpot <sup>4</sup> | | X | | | | | | | | | | | | | | | | X | | |
| Blood<br>collection for<br>research<br>sample <sup>4,15</sup> | | X | | | | X | X | | | | X | X | X | | | | X | X | X | X |
| HLA typing<br>(optional) | | | | | | | | | | | | | | | | | | | X <sup>19</sup> | X <sup>19</sup> |
| Laser imaging<br>and capsaicin<br>challenge <sup>4</sup> | X | X | | | | | X | | | | | X | X | | | | | X | X <sup>16</sup> | X <sup>16</sup> |

Abbreviations: AE = adverse event; CRU = Clinical Research Unit; D = day; DBF = dermal blood flow; ECG = electrocardiogram; EoS = End of Study; EoT = End of Treatment; ET = Early Termination; FSH = follicle-stimulating hormone; H = hour; HBV = hepatitis B virus; HCV = hepatitis C virus; HIV = human immunodeficiency virus; IM = intramuscular; IMP = investigational medicinal product; LSCI = Laser Speckle Contrast Imaging; MRI = magnetic resonance imaging; PBMC = peripheral blood mononuclear cell; PD = pharmacodynamic; SAE = serious adverse event; SD = standard deviation; SRN = Screening; TC = telephone call, V = visit

- 1. The Investigator may perform visits outside of the scheduled study visits (unscheduled visits) listed in the table to conduct evaluations or assessments required to protect the well-being of the participant.
- 2. Screening and V1 visits can be rescheduled, and Screening window may be extended.
- 3. AEs/SAEs recording from time of informed consent up to and including Follow-up or ET.
- 4. On IMP administration days, all laboratory, PD, and capsaicin assessments are to be performed prior to IMP administration.
- 5. After each IMP administration, (a) participants will stay for 6 hours (±2 hours) after injection for safety observation (except for sentinel participants who will stay for 24 hours after the first dose), (b) participants (except the sentinels' first dose) will have an approximately 24-hour onsite safety review including review of vital signs, temperature, diary, AEs, and medications, (c) all participants will have a telephone call approximately 48-hours post IMP injection for safety check including AE and medication review, and (d) all participants will complete a diary daily for 7 days, starting from the day of IMP administration.
- 6. On IMP administration days, vital signs (including temperature) will be measured before and after IMP administration.
- 7. Participants should be resting in a semi-recumbent position for at least 10 minutes before vital signs measurements. Semi-recumbent vital signs will include heart rate, systolic and diastolic blood pressure, respiratory rate, and body temperature.
- 8. Full neurological and physical examinations are to be performed during Screening, at Week 16 (EoT), Week 44 (EoS), and ET; brief (targeted) examinations may be performed at all other visits.
- 9. Laboratory assessments are detailed in Section 7.7 and Appendix 1.



#### Clinical Trial Protocol

- 10. A diary will be dispensed on Day 1. Participants will complete it for 7 days daily, starting on the day of each administration of IMP.
- 11. For females of childbearing potential only, blood pregnancy test at Screening and urine test at other visits. For females of nonchildbearing potential in post-menopausal state, FSH at screening.
- 12. Inflammatory measures in blood will include but are not limited to C-reactive protein and erythrocyte sedimentation rate. At Screening only, antinuclear antibody, IgM rheumatoid factor, and anti-cyclic citrullinated peptide.
- 13. Cytokine blood samples will be collected pre-dose and approximately 6 hours (±2 hours) post-dose, and only analyzed at the Investigator's discretion if clinically indicated; otherwise, they will be analyzed at the EoT visit. The cytokine panel will include but is not limited to IFN-γ, IL-2, IL-4, IL-6, IL-8, and TNF-α.
- 14. Antibody measures in blood, including but not limited to anti-CGRP target epitope, anti-UBITh, anti-CpG1, and isotyping of anti-CGRP antibodies.
- 15. A sample to be obtained as allowed by local regulations and participant consent.
- 16. After Week 16, LSCI assessment may no longer be required once the average capsaicin-induced DBF increase within that cohort has returned to baseline (i.e., DBF response ±2 SD before administration of IMP within a cohort).
- 17. Historic MRI within 90 days of Screening may be accepted.
- 18. IMP should be administered to the opposite arm that was used to take blood. Alternate arms should be used for injection visits and the arm used for IMP administration should be
- 19. A blood sample to be obtained for HLA typing at any post-Week 16 visit as allowed by participant consent. Blood sample is only to be collected at one visit.